CLINICAL TRIAL: NCT02935985
Title: Emergency Management of Spontaneous Intracerebral Haemorrhage - Biomarkers
Acronym: EsICH
Status: Completed | Type: Observational
Sponsor: Iuliu Hatieganu University of Medicine and Pharmacy (Other)
Responsible Party: Principal Investigator, Eugenia-Maria Muresan, Coordinating Investigator, Iuliu Hatieganu University of Medicine and Pharmacy
Other Study IDs: 21288/ 04.10.2016
Record Dates: First submitted 2016-10-14; First posted 2016-10-18 (Estimated); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Cerebral Hemorrhage
Keywords: spontaneous intracerebral hemorrhage; point-of-care bio-markers; multicenter; Emergency Department; Romania
MeSH Terms: conditions — Cerebral Hemorrhage; Emergencies | interventions — C-Reactive Protein; fibrin fragment D; Blood Cell Count; Glucose; Cholesterol; Cholesterol, LDL; Triglycerides; Fibrinogen

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Venous blood samples will be collected from patients who have suffered a spontaneous intracerebral hemorrhage less than 8h ago.
  Point-of-care bio-markers will be assessed by using an immunoanalyzer in the Emergency Department.
  From the blood samples used for determining the other biological parameters (CBC, biochemistry, coagulogram).
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Adults with sICH less than 8h: Adult patients presenting in one of the study locations and being diagnosed with intracerebral hemorrhage. The onset of the conditions is establised as sonner than 8h.
  Clinical evaluations will be performed, along with collecting venous blood samples for determining point-of-care bio-markers and biological parameters.
  Participants will be assessed (clinically or by telephone) over a period of 180 days.
  Interventions: Other: Point-of-care bio-markers (cTnI, hsCRP, D-Dimer) and biological parameters (CBC, glucose, cholesterol, LDL cholesterol, triglycerides, fibrinogen)

INTERVENTIONS:
Other: Point-of-care bio-markers (cTnI, hsCRP, D-Dimer) and biological parameters (CBC, glucose, cholesterol, LDL cholesterol, triglycerides, fibrinogen) — Clinical evaluations will be performed, along with collecting venous blood samples for determining point-of-care bio-markers and biological parameters.
  Participants will be assessed (clinically or by telephone) over a period of 180 days.

SUMMARY:
The bio-markers substudy of EsICH is designed to recruit patients with acute (first 8h) spontaneous intracerebral hemorrhage and assess a series of biological parameters (CBC, glucose, cholesterol, LDL cholesterol, triglycerides) and point-of-care bio-markers (cTnI, hsCRP, D-Dimer) in order to predict the functional outcome of these patients and to determine their input for early risk stratification and prognosis.

DETAILED DESCRIPTION:
EsICH is designed as a multicenter double blind randomized (2:1) clinical trial assessing the effects of tranexamic acid (2g in total) on patients with acute (first 8h) spontaneous intracerebral hemorrhage.

The bio-markers substudy addresses the same category of patients and assesses biological parameters (CBC, glucose, cholesterol, LDL cholesterol, triglycerides) and point-of-care bio-markers (cTnI, hsCRP, D-Dimer) in order to predict the functional outcome of these patients and to determine their input for early risk stratification and prognosis.

The patients with a diagnostic CT scan are recruited in the Emergency Departments or Neurology/ Neurosurgery Wards of the hospitals enrolled in the study and blood samples are drawn in the first 8h from the onset of the condition. The patient is then clinically assessed by the study investigators for the first 7 days of the admission and a second CT scan is performed on the second day (24h from the onset of the condition).

Telephone follow-ups will be completed on day 90 and 180 by the coordinating center of the study.

The bio-markers substudy is an observational, prospective multicenter (the study will be initially started in one center - Cluj-Napoca - and then the Tirgu Mures center will be activated. Two more centers might be also included on a later time - Alba and Bistrita-Nasaud, pending on financial and logistic reasons).

ELIGIBILITY:
Inclusion Criteria:

1. Age over 18 years old
2. CT scan diagnosis of an spontaneous intracerebral hemorrhage in the first 8h from the onset of the condition
3. Informed consent
4. Access to telephone evaluations (landline or mobile phone for the participant or a family member)

Exclusion Criteria:

1. GCS < 8 points
2. Secondary cause of the intracerebral hemorrhage (trauma, known AVM, aneurysm, hemorrhagic transformation of an ischemic stroke, thrombosis of central veins and sinuses, thrombolitic therapy, tumors, infections).
3. Severe disability prior to this hemorrhagic event (modified Rankin Score =>4);
4. Known venous thrombembolic condition
5. History of coagulopathy (genetic or acquired)
6. Recent ischemic events (< 12 months) (ischemic stroke, myocardial infarction, peripheric artheriopathy)
7. History of seizures (or present condition)
8. Undergoing treatment with heparin, LMWH, GPIIb/IIIa antagonists or oral anticoagulants (warfarin/ acenocumarol, factor Xa inhibitors, thrombin inhibitors - in the last 14 days)
9. Pregnancy or breast feeding
10. Scheduled neurosurgical intervention on the next 24h
11. Ongoing of scheduled hemostatic treatment - prothrombin, vitamin K, fresh frozen plasma, platelets
12. Enrollment in other clinical trials in the last 30 days
13. Known terminal stage disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients presenting in one of the study centers and having a diagnostic CT scan for intracerebral hemorrhage less than 8h old.
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2016-12-12 (Actual); Primary Completion 2018-06-11 (Actual); Study Completion 2018-11-24 (Actual)

PRIMARY OUTCOMES:
Assessment of the correlation between point-of-care bio-markers (cTnI, hsCRP, D-Dimer) and biological parameters (CBC, glucose, cholesterol, LDL cholesterol, triglycerides, fibrinogen) and the functional recovery of SICH patients on day 180. | 180 days from the enrollment
  Functional outcomes are defined as modified Rankin Score of 0 to 3 and Barthel Index of 60 to 100 points.

SECONDARY OUTCOMES:
Assessment of the correlation between point-of-care bio-markers (cTnI, hsCRP, D-Dimer) and biological parameters (CBC, glucose, cholesterol, LDL cholesterol, triglycerides, fibrinogen) and the hematoma volume. | 2 days from the enrollment
Assessment of the correlation between point-of-care bio-markers (cTnI, hsCRP, D-Dimer) and biological parameters (CBC, glucose, cholesterol, LDL cholesterol, triglycerides, fibrinogen) and the edema surrounding the bleeding site | 2 days from the enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Eugenia M Muresan, MD, PhD stud, Principal Investigator — Iuliu Hatieganu University of Medicine and Pharmacy Cluj-Napoca
Locations (2):
- Romania (2):
  - Emergency Clinical County Hospital Cluj-Napoca - Emergency Department, Cluj-Napoca, Cluj
  - Emergency Clinical County Hospital Cluj-Napoca - Neurology ward, Cluj-Napoca, Cluj

IPD SHARING:
Plan to Share IPD: No